CLINICAL TRIAL: NCT03807986
Title: The Combination Therapy of Nanofat Grafting and Platelet-Rich Plasma Injection Compared With Microfat Grafting and Platelet-Rich Plasma Injection Synergy in Treating Striae Distensae
Brief Title: The Combination Therapy of Nanofat Grafting and PRP Compared With Microfat Grafting and PRP Synergy in Treating Striae Distensae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Jinan University (Other)
Collaborators: Science and Technology Program of Guangzhou,Guangzhou Sipintang Biological technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Li-Ling Xiao, Associate Chief of Department of Plastic Surgery, First Affiliated Hospital of Jinan University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Xiao FirstJinanU
Record Dates: First submitted 2019-01-02; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Treatments of Striae Distensae
Keywords: Striae Distensae; Platelet-Rich Plasma (PRP); Nanofat Graft; Microfat Graft; Combination Therapy
MeSH Terms: conditions — Striae Distensae | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanofat grafting and PRP injection (Experimental): Striae diatensae will be treated by nanofat grafting once every three months for 2 times combined with PRP injection once a month for 6 times.
  Interventions: Procedure: Nanofat grafting; Procedure: Platelet-rich plasma (PRP) Injection
- Microfat grafting and PRP injection (Experimental): Striae diatensae will be treated by microfat grafting once every three months for 2 times combined with PRP injection once a month for 6 times.
  Interventions: Procedure: Microfat grafting; Procedure: Platelet-rich plasma (PRP) Injection

INTERVENTIONS:
Procedure: Nanofat grafting — Nanofat grafting will be applied once every three months for 2 times.
  Arms: Nanofat grafting and PRP injection
Procedure: Microfat grafting — Microfat grafting will be applied once every three months for 2 times.
  Arms: Microfat grafting and PRP injection
Procedure: Platelet-rich plasma (PRP) Injection — PRP Injection will be applied once a month for 6 times.

SUMMARY:
Striae distensae is caused by the fracture and damage of the elastic fibers and collagen fibers, which is still a difficulty to overcome. Based on the studies demonstrated that platelet-rich plasma(PRP) has positive effect on superficial scar, and nanofat and microfat are effective in treating atrophic scar. So in this clinical trial, the investigators are going to treat striae distensae by using two combination therapies. One is nanofat grafting and PRP injection synergy, and the other one is treated by microfat grafting with PRP injection.

DETAILED DESCRIPTION:
The participants were randomly assigned into two groups. Group A is treated by nanofat grafting once every three months for 2 times combined with PRP injection once a month for 6 times. Group B will be treated by microfat grafting onceevery three months for 2 times combined with PRP injection once a month for 6 times. The participants were asked to come back 1、3、6、9 months after treatment for further follow-up.Before and after the treatment, the striae distensae will be assessed subjectively by satisfaction assessment, and objectively by ultrasound and immunohistochemical analysis.

ELIGIBILITY:
Inclusion Criteria:

* The striae distensae
* Age ≤ 35 years old

Exclusion Criteria:

* Skin allergy
* Cicatricial diathesis
* Skin inflammation or wound
* Platelet dysfunction syndrome
* Take anticoagulant drugs
* Acute or chronic infection
* Chronic liver disease
* Active vitiligo, psoriasis, systemic lupus erythematosus

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemical analysis | Change from baseline at 15 months.
  The tissue extracted will be taken for immunohistochemical analysis to observe the amount of elastic fiber and collagen fiber,etc. More collagen fiber generated better outcome of the treatments.

SECONDARY OUTCOMES:
Ultrasound | Change from baseline dermal thickness at 3,6,9,12,15 months of the treatments.
  The striae distensae will be assessed by ultrasound in order to observe the change of dermal thickness of striae after the application of nanofat or microfat grafting with PRP injection. if the treatments worked, the dermal thickness will be increased.
Ultrasound | Change from baseline width of striae at 3,6,9,12,15 months of the treatments.
  The striae distensae will be assessed by ultrasound in order to observe the change of width of striae after the application of nanofat or microfat grafting with PRP injection. Smaller the width better the results.

OTHER OUTCOMES:
Satisfaction assessments of participants: questionnaire | At 15th month.
  The participants will fill in a questionnaire about the efficacy of the treatments. Participants will choose one of the following answers 'satisfied, unchanged, not satisfied' as feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Li Ling Xiao, MD, Principal Investigator — First Affiliated Hospital of Jinan University
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson RE, Parry EJ, Humphries JD, Jones CJ, Polson DW, Kielty CM, Griffiths CE. Fibrillin microfibrils are reduced in skin exhibiting striae distensae. Br J Dermatol. 1998 Jun;138(6):931-7. doi: 10.1046/j.1365-2133.1998.02257.x. PMID 9747352
- [Background] Cho C, Cho E, Kim N, Shin J, Woo S, Lee J, Lee J, Lee E, Ha J. Biophysical properties of striae rubra and striae alba in human skin: Comparison with normal skin. Skin Res Technol. 2019 May;25(3):283-288. doi: 10.1111/srt.12645. Epub 2018 Oct 22. PMID 30345576
- [Background] Forbat E, Al-Niaimi F. Treatment of striae distensae: An evidence-based approach. J Cosmet Laser Ther. 2019;21(1):49-57. doi: 10.1080/14764172.2017.1418515. Epub 2018 Feb 16. PMID 29451986
- [Background] Hague A, Bayat A. Therapeutic targets in the management of striae distensae: A systematic review. J Am Acad Dermatol. 2017 Sep;77(3):559-568.e18. doi: 10.1016/j.jaad.2017.02.048. Epub 2017 May 24. PMID 28551068

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03807986/Prot_SAP_000.pdf